CLINICAL TRIAL: NCT05687370
Title: Modified Dynamic Needle Tip Positioning Versus Long-Axis In-Plane Ultrasound Guided Radial Artery Cannulation in Patients With Coronary Artery Disease: A Randomized Controlled Trial
Brief Title: Modified Dynamic Needle Tip Positioning vs Conventional Long-axis In-plane in Radial Artery Cannulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Meng Lv, Professor, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: YXLL-KY-2022(104)
Record Dates: First submitted 2022-12-04; First posted 2023-01-18 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Ultrasound; Arterial Catheterization; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified dynamic needle tip positioning technique (Active Comparator): In Modified dynamic needle tip positioning technique, short-axis in-plane is used, needle tip was dynamic guided by ultrasound that added two developing lines on the ultrasonic probe.
  Interventions: Procedure: Modified dynamic needle tip positioning under ultrasound-guidance
- Long-axis in-plane technique (Active Comparator)
  Interventions: Procedure: Long-axis technique

INTERVENTIONS:
Procedure: Modified dynamic needle tip positioning under ultrasound-guidance — The tip of needle is positioned under ultrasound-guidance using modified dynamic short-axis view.
  Arms: Modified dynamic needle tip positioning technique
Procedure: Long-axis technique — The tip of needle is positioned under ultrasound-guidance using conventional long-axis in-plane view.
  Arms: Long-axis in-plane technique

SUMMARY:
Conventionally, long-axis in-plane (LA-IP), short-axis out-of-plane (SA-OOP) and dynamic needle tip positioning based on SA-OOP views are commonly used method to image the target vessel during cannulation under US guidance. A modified SA-OOP that add developing line on the ultrasonic probe improve the success rate of cannula insertion into the radial artery on the first attempt.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnostic criteria of coronary atherosclerotic heart disease according to the tenth version of international Classification of diseases(ICD-10);
2. Requires invasive arterial blood pressure monitoring;
3. New York Heart Association(NYHA) classification I, II or III;
4. The American Society of Anesthesiologists (ASA) classification I, II or III;
5. Patients older than 18 years and younger than 85 years (Adult);
6. Patients signed the informed consent before the study.

Exclusion Criteria:

1. Patients with hemodynamically unstable (systolic blood pressure 60 or less);
2. Patients with abnormal results of the modified Allen test;
3. Patients with ulnar artery occlusion;
4. Patients with coagulation disorders;
5. Patients with skin abnormalities such as inflammation or hematoma at the cannulation site;
6. Patients with raynaud disease and prevalent atherosclerosis;
7. Patients with history of hand or wrist trauma or surgery;
8. Patients who have undergone radial artery interventional therapy or radial artery cannulation within 3 months on the puncture side;
9. Patients with BMI more than 40 kg/m2;
10. Patients who have participated in other relevant clinical studies within 3 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-03-26 (Actual); Study Completion 2023-03-26 (Actual)

PRIMARY OUTCOMES:
Success rate of the radial artery cannulation at first attempt | intraoperative
  Successful confirmation of the arterial waveform through a pressure monitor at first attempt of the radial artery cannulation

SECONDARY OUTCOMES:
Time of arterial catheterization | Interval between contact of the ultrasound transducer with the skin and confirmation of an arterial waveform on the monitor, an expected average observation time of 300 seconds
Time to first puncture of the artery | Interval between skin penetration of the needle and flashback of blood, an expected average of 200 seconds
Time ultrasound imaging | Interval between contact of the ultrasound transducer with the skin and penetration of the needle through the skin, , an expected average of 100 seconds
Number of puncture attempts | Up to 5 times, an expected average observation time of 70 seconds
Vascular complications in the surgery | postoperative, within 24 hours
  including thrombosis, hematoma, and vasospasm

CONTACTS AND LOCATIONS:
Overall Officials: Meng Lv, doctor, Principal Investigator — Jinan, Shandong Province, China, 250000
Locations (1):
- Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No